CLINICAL TRIAL: NCT02663440
Title: Trial of Hypofractionated Intensity Modulated Radiation Therapy With Temozolomide and Granulocyte-macrophage Colony-stimulating Factor for Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZJZLYY-HN-2016-01
Record Dates: First submitted 2016-01-18; First posted 2016-01-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Temozolomide

ARMS (1):
- IMRT (Experimental): Hypofractionated IMRT With Temozolomide and Granulocyte-macrophage Colony-stimulating Factor
  Interventions: Radiation: Hypofractionated IMRT; Biological: Granulocyte-macrophage Colony-stimulating Factor; Drug: Temozolomide

INTERVENTIONS:
Radiation: Hypofractionated IMRT — Hypofractionated IMRT
Biological: Granulocyte-macrophage Colony-stimulating Factor — Granulocyte-macrophage Colony-stimulating Factor
Drug: Temozolomide — Temozolomide

SUMMARY:
Phase II Trial of Hypofractionated Intensity Modulated Radiation Therapy(IMRT) With Temozolomide and Granulocyte-macrophage Colony-stimulating Factor(GM-CSF) for Patients With Newly Diagnosed Glioblastoma Multiforme.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed and pathologically confirmed glioblastoma multiforme without an enhanced lesion beside the cerebrospinal fluid space on baseline magnetic resonance imaging
* Karnofsky performance status more than 60
* Normal liver, kidney, and bone marrow function.

Exclusion Criteria:

* Previous allergies to granulocyte macrophage colony stimulating factor
* Receiving radiotherapy
* Receiving other investigational agents
* Had uncontrolled intercurrent illnesses.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Cao C, Wang L, Jiang F, Jin Q, Jin T, Huang S, Hu Q, Chen Y, Piao Y, Hua Y, Feng X, Zhou Y, Chen X. Granulocyte-macrophage colony-stimulating factor for newly diagnosed glioblastoma. Neoplasia. 2025 May;63:101156. doi: 10.1016/j.neo.2025.101156. Epub 2025 Mar 15. PMID 40090128